CLINICAL TRIAL: NCT02162433
Title: Does Dexmedetomidine Decrease the Incidence of Untoward Airway Events After Deep or Awake Extubation in Patients Undergoing Adenotonsillectomy With or Without Myringotomy and Tube Placement?
Brief Title: The Effect of Dexmedetomidine on Airway Complications After Deep or Awake Extubation
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Terminated due to a high number of protocol deviations secondary to non-study approved opioid administration.
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Principal Investigator, Makara Cayer, Prinicpal Investigator, Massachusetts Eye and Ear Infirmary
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 14-019H
Record Dates: First submitted 2014-06-10; First posted 2014-06-12 (Estimated); Results first posted 2020-04-09 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Adenotonsillar Hypertrophy; Obstructive Sleep Apnea; Tonsillitis; Adenoiditis
MeSH Terms: conditions — Sleep Apnea, Obstructive; Tonsillitis | interventions — Saline Solution; Sodium Chloride; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1. Awake extubation/dexmedetomidine (Active Comparator): Awake extubation receiving dexmedetomidine.
  Interventions: Drug: Dexmedetomidine
- 2. Awake extubation/placebo (Placebo Comparator): Awake extubation receiving placebo (normal saline).
  Interventions: Drug: Normal Saline
- 3.Deep extubation/dexmedetomidine (Active Comparator): Deep extubation receiving dexmedetomidine.
  Interventions: Drug: Dexmedetomidine
- 4. Deep extubation/placebo (Placebo Comparator): Deep extubation receiving placebo (normal saline).
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Normal Saline — to arms 2,4. Serves as the placebo.
  Other Names: 0.9% Sodium Chloride Solution
  Arms: 2. Awake extubation/placebo; 4. Deep extubation/placebo
Drug: Dexmedetomidine — to arms 1,3
  Other Names: Precedex
  Arms: 1. Awake extubation/dexmedetomidine; 3.Deep extubation/dexmedetomidine

SUMMARY:
The investigators aim to investigate the effect of dexmedetomidine on the perioperative respiratory complications in this patient population undergoing both awake and deep tracheal extubation.

DETAILED DESCRIPTION:
We propose a prospective double-blinded randomized controlled trial. 336 pediatric patients presenting to Massachusetts Eye and Ear Infirmary (MEEI) for adenotonsillectomy who are eligible for the study based on inclusion and exclusion criteria will be recruited. A Clinical Pharmacy specialist, will be in charge of preparing the dexmedetomidine and placebo doses and will randomize the patients to four equally numbered groups. The anesthesiologist will receive the assignment for the extubation method in a sealed envelope from the Clinical Pharmacy specialist. Multiple parameters will be recorded in perioperative period to quantify perioperative adverse respiratory events.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 3 to 16 years of age undergoing adenotonsillectomy, with or without myringotomy or myringoplasty
* ASA 1 & 2

Exclusion Criteria:

* Known allergy or hypersensitivity reaction to dexmedetomidine
* Organ dysfunction (renal/hepatic failure or leukemia)
* Cardiac disease (congenital or acquired)
* Airway or thoracic malformation
* Cerebral palsy
* Hypotonia
* Need for premedication
* Current/recent upper respiratory infection (within four weeks prior to the surgery)
* Asthma
* Allergy or intolerance to clonidine
* Non-English speaking parents/patients.

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 92 (Actual)
Dates: Start 2015-03; Primary Completion 2018-04 (Actual); Study Completion 2018-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Makara Cayer, MD, Principal Investigator — MEEI/ Harvard Medical School
Locations (1):
- MEEI, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1. Awake Extubation/Dexmedetomidine | 2. Awake Extubation/Placebo | 3.Deep Extubation/Dexmedetomidine | 4. Deep Extubation/Placebo
Started | 23 | 23 | 23 | 23
Completed | 22 | 21 | 21 | 22
Not Completed | 1 | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1. Awake Extubation/Dexmedetomidine | 2. Awake Extubation/Placebo | 3.Deep Extubation/Dexmedetomidine | 4. Deep Extubation/Placebo | Total
Number analyzed (Participants) | 23 | 23 | 23 | 23 | 92
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 23 | 23 | 23 | 23 | 92
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.64 (3.21) | 6.1 (2.89) | 6.52 (2.79) | 6.64 (2.8) | 6.48 (2.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 12 | 9 | 39
  Male | 14 | 14 | 11 | 14 | 53
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 23 | 23 | 23 | 23 | 92

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Respiratory Complications
Description: Number of patients exhibiting any of the following outcomes:
  1. desaturation to less than 95% for more than 10 seconds;
  2. breath holding;
  3. complete or partial laryngospasm;
  4. bronchospasm;
  5. croup;
  6. number of episodes of persistent cough (three or more consecutive coughs);
  7. negative pressure pulmonary edema;
  8. stridor.
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | 1. Awake Extubation/Dexmedetomidine | 2. Awake Extubation/Placebo | 3.Deep Extubation/Dexmedetomidine | 4. Deep Extubation/Placebo
Number analyzed (Participants) | 22 | 21 | 21 | 22
Participants | 13 | 15 | 13 | 17

2. Secondary Outcome: Number of Participants With Emergence Agitation
Description: Number of patients with an incidence of emergence agitation post-surgery defined by the Pediatric Anesthesia Emergence Delirium (PAED) scale of >10.
  Emergence agitation is characterized by non-purposeful movement, restlessness, thrashing, incoherence, inconsolability, and unresponsiveness. The PAED is a scale used to assess emergence agitation in our patient population. It's minimum value is zero and maximum value is 20, with 0 being no emergence agitation and 20 being the most agitated state.
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | 1. Awake Extubation/Dexmedetomidine | 2. Awake Extubation/Placebo | 3.Deep Extubation/Dexmedetomidine | 4. Deep Extubation/Placebo
Number analyzed (Participants) | 22 | 21 | 21 | 22
Participants | 7 | 13 | 9 | 13

3. Secondary Outcome: Number of Participants With Postoperative Nausea and Vomiting (PONV)
Description: Number of patients who experienced postoperative nausea and vomiting (PONV) as noted by the parental questionnaire administered 24 hours after the patient is discharged.
Time Frame: 24 hrs
Measure: Count of Participants; unit: Participants
Arm/Group | 1. Awake Extubation/Dexmedetomidine | 2. Awake Extubation/Placebo | 3.Deep Extubation/Dexmedetomidine | 4. Deep Extubation/Placebo
Number analyzed (Participants) | 22 | 21 | 21 | 22
Participants | 5 | 6 | 6 | 3

4. Secondary Outcome: Average Time From End of Surgery to Leaving the Operating Room
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | 1. Awake Extubation/Dexmedetomidine | 2. Awake Extubation/Placebo | 3.Deep Extubation/Dexmedetomidine | 4. Deep Extubation/Placebo
Number analyzed (Participants) | 22 | 21 | 21 | 22
Minutes | 19.15 (5.5) | 18.05 (7.43) | 10.29 (3.73) | 11.77 (5.6)

5. Secondary Outcome: The Average Time From Admission to the PACU to Discharge Home (Excluding Overnight Admission)
Time Frame: 24 hrs
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | 1. Awake Extubation/Dexmedetomidine | 2. Awake Extubation/Placebo | 3.Deep Extubation/Dexmedetomidine | 4. Deep Extubation/Placebo
Number analyzed (Participants) | 22 | 21 | 21 | 22
Minutes | 345.06 (91.23) | 320.19 (69.07) | 341.53 (73.85) | 328.05 (93.97)

6. Secondary Outcome: Number of Participants Needing Follow-up Pain Medication
Description: 24-hour postoperative pain medication requirement assessed by a parental questionnaire administered 24 hours after discharge. The parents are asked whether their child took any pain medication within the last 24 hours since the surgery.
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | 1. Awake Extubation/Dexmedetomidine | 2. Awake Extubation/Placebo | 3.Deep Extubation/Dexmedetomidine | 4. Deep Extubation/Placebo
Number analyzed (Participants) | 22 | 21 | 21 | 22
Participants | 18 | 17 | 20 | 18

7. Secondary Outcome: Number of Patients With Unplanned Hospital Admission
Description: Any unplanned hospital admission due to perioperative respiratory adverse events.
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | 1. Awake Extubation/Dexmedetomidine | 2. Awake Extubation/Placebo | 3.Deep Extubation/Dexmedetomidine | 4. Deep Extubation/Placebo
Number analyzed (Participants) | 22 | 21 | 21 | 22
Participants | 0 | 2 | 0 | 0

ADVERSE EVENTS:
Time Frame: 24 hours post-op
Arm/Group | 1. Awake Extubation/Dexmedetomidine | 2. Awake Extubation/Placebo | 3.Deep Extubation/Dexmedetomidine | 4. Deep Extubation/Placebo
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/21 | 0/21 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/21 | 0/21 | 0/22
Other Adverse Events (participants affected / at risk) | 13/22 | 15/21 | 13/21 | 17/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1. Awake Extubation/Dexmedetomidine (N=22) | 2. Awake Extubation/Placebo (N=21) | 3.Deep Extubation/Dexmedetomidine (N=21) | 4. Deep Extubation/Placebo (N=22)
Post-extubation persistent cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 6 (6) | 1 (1) | 4 (4)
PACU persistent cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5) | 8 (8) | 9 (9)
Post-extubation low SaO2 (Blood and lymphatic system disorders) | 6 (6) | 4 (4) | 0 (0) | 1 (1)
PACU low SaO2 (Blood and lymphatic system disorders) | 6 (6) | 6 (6) | 8 (8) | 7 (7)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nausea/Vomiting (General disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Post-Extubation Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
PACU stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Post-Extubation Croup (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
PACU Croup (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Post-Extubation Breath Holding (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
PACU Breath Holding (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Tonsil Bleed (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Informed Consent Form (2018-01-29): https://cdn.clinicaltrials.gov/large-docs/33/NCT02162433/ICF_000.pdf
  • Study Protocol (2018-01-29): https://cdn.clinicaltrials.gov/large-docs/33/NCT02162433/Prot_001.pdf
  • Statistical Analysis Plan (2020-02-07): https://cdn.clinicaltrials.gov/large-docs/33/NCT02162433/SAP_002.pdf